CLINICAL TRIAL: NCT04475198
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ST-2427 IV Infusion in Healthy Subjects
Brief Title: Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ST-2427
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: strategic decision
Sponsor: SiteOne Therapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST-2427-CS-001; 1UG3DA049599 (NIH)
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Acute, Post-operative Pain
Keywords: Pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single Ascending Dose: Cohort 1 (Experimental): 5 mg ST-2427 (n=4) or placebo (n=2) administered once over a 60-minute intravenous (IV) infusion. 2 sentinel subjects will receive dosing for review of safety data (ST-2427 n=1, placebo n=1) before remainder of cohort.
  Interventions: Drug: ST-2427; Drug: Placebo
- Single Ascending Dose: Cohort 2 (Experimental): 10 mg ST-2427 (n=4) or placebo (n=2) administered once over a 60-minute intravenous (IV) infusion.
  Interventions: Drug: ST-2427; Drug: Placebo
- Single Ascending Dose: Cohort 3 (Experimental): 15 mg ST-2427 (n=4) or placebo (n=2) administered once over a 60-minute intravenous (IV) infusion.
  Interventions: Drug: ST-2427; Drug: Placebo
- Single Ascending Dose: Cohort 4 (Experimental): 22 mg ST-2427 (n=4) or placebo (n=2) administered once over a 60-minute intravenous (IV) infusion.
  Interventions: Drug: ST-2427; Drug: Placebo
- Single Ascending Dose: Cohort 5 (Experimental): 33 mg ST-2427 (n=4) or placebo (n=2) administered once over a 60-minute intravenous (IV) infusion.
  Interventions: Drug: ST-2427; Drug: Placebo

INTERVENTIONS:
Drug: ST-2427 — Investigational drug
Drug: Placebo — 5% Dextrose Injection

SUMMARY:
This randomized, double-blind, placebo controlled, study will be conducted to evaluate the safety, tolerability, and pharmacokinetics of ST-2427. Subjects will be randomized to receive a single dose of ST-2427 or placebo in a Single Ascending Dose (SAD) design.

A total of 30 subjects will be enrolled. Subjects will be randomized in a 4:2 ratio of ST-2427 to placebo. Study drug will be blinded to all subjects and investigators.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled study in healthy adult males and females of non-child-bearing potential to evaluate the safety, tolerability, and pharmacokinetics (PK) of ST-2427. This trial will include careful assessments of treatment effects on vital signs including cardiac and respiratory function and body temperature over a range of doses of ST-2427, administered as single doses. SiteOne Therapeutics, Inc. plans to use the safety, tolerability, and PK findings from this study to inform the doses and study design for Phase 2 clinical studies in subjects with acute post-operative pain.

Approximately 30 subjects, 6 subjects into each of 5 cohorts, will be enrolled in this study at a single clinical site.

Subjects will be randomized 4:2 to receive a single dose of ST-2427 or placebo in a Single Ascending Dose (SAD) design. The Study will evaluate 5 dose strengths of ST-2427, one dose level in each of 5 cohorts of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who meet the following criteria will be eligible for inclusion:

  1. Healthy adult males and/or females (of non-childbearing potential), 18 to 55 years of age (inclusive) at the time of screening;
  2. Body mass index (BMI) within 18.0 to 35.0 kg/m2, inclusive (minimum weight of at least 50.0 kg at Screening);
  3. Medically healthy without clinically significant abnormalities at the screening visit, including physical examination and vital signs within the following ranges: heart rate 50 to 100 bpm, systolic blood pressure 100 to 149 mmHg; diastolic 70 to 94 mmHg;
  4. The mean QTcF interval duration ≤450 msec for males and ≤470 msec for females measured from the triplicate ECGs taken at least 1 minute apart with QT wave corrected for heart rate (HR) using Fredericia's method
  5. Hemoglobin/hematocrit, white blood cell (WBC) count, and platelet count equal to or greater than the lower limit of normal range of the reference laboratory (may be confirmed upon repeat testing without Sponsor approval);
  6. Creatinine, blood urea nitrogen (BUN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal to or less than the upper limit of normal for the reference laboratory (may be confirmed upon repeat testing); results of all other clinical chemistry and urine analytes without any clinically significant abnormality;
  7. Non-smokers (including tobacco, e-cigarettes or marijuana), and no use of any tobacco product for at least 1 month prior to admission in the study;
  8. Willing and able to provide written informed consent;
  9. Willing and able to comply with all study assessments and adhere to the protocol schedule;
  10. Have suitable venous access for blood sampling, as determined by an Investigator at screening;
  11. If female, be of non-childbearing potential (e.g. post-menopausal as demonstrated by follicle stimulating hormone (>40 mIU/mL), or surgically sterilized by tubal ligation or hysterectomy). Site personnel's review of the subject's medical records, medical examination, or medical history interview is acceptable evidence of female sterilization, verbal confirmation is adequate;
  12. If male, willing not to donate sperm from the time of first study drug administration until 90 days after the final administration of study drug. If male and not intending to engage in sexual intercourse over the duration of the study, willing to agree to abstinence at screening. If male and engaging in sexual intercourse, willing to use a double barrier method of contraception (condom and spermicide). The latter criterion applies to all males (and/or female partners) including males who are surgically sterile and must be followed from the time of first study drug administration until 90 days after the final administration of study drug.

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any of the following criteria:

  1. History or presence of significant cardiovascular (including arrhythmia and ventricular tachyphylaxis), pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by an Investigator to be clinically relevant;
  2. Creatinine, blood urea nitrogen (BUN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal to 1.5 x upper limit of normal for the reference laboratory (may be confirmed upon repeat testing);
  3. History of orthostatic reactions
  4. Orthostatic reaction at screening defined as drop in systolic blood pressure by ≥20 mmHg or drop in systolic blood pressure to <90 mmHg on standing for 3 minutes from the supine position.
  5. History of seizure disorders, except for non-complex febrile seizures in childhood with absence of non-febrile seizures in parents and siblings.;
  6. Positive urine drug/alcohol testing at Screening or Day -2;
  7. Positive test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Antibody (HCVAb);
  8. Positive test results for COVID-19 (PCR or Antibodies)
  9. History of substance abuse or alcohol abuse (defined as greater than 2 standard drinks per day) within the previous 2 years;
  10. Use of any prescription medication or any over-the-counter medication, including herbal products and vitamins within 14 days or 5 half-lives (whichever is longer) prior to randomization;
  11. Documented hypersensitivity reaction or anaphylaxis to any medication;
  12. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening, or receipt of a blood transfusion within 1 year of screening;
  13. Dosed in another investigational clinical trial within 30 days prior to Screening;
  14. Any condition or prior therapy, e.g. seizures, or head trauma, that may lead to CNS effects during the study;
  15. Documented or self-reported history of orthostatic hypotension or symptoms of hypotension such as dizziness, syncope or blurred vision upon standing;
  16. Any condition which is associated with increased brain permeability, e.g. cerebral ischemia, brain trauma, multiple sclerosis, brain tumors, brain infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Jerling, MD, PhD, Study Director — Unaffliated
Locations (1):
- Altasciences, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Ascending Dose: Cohort 1: 5 mg ST-2427 (n=4) administered once over a 60-minute intravenous (IV) infusion.
  ST-2427: Investigational drug
- Single Ascending Dose: Cohort 2: 10 mg ST-2427 (n=4) administered once over a 60-minute intravenous (IV) infusion.
  ST-2427: Investigational drug
- Single Ascending Dose: Cohort 3: 15 mg ST-2427 (n=4) administered once over a 60-minute intravenous (IV) infusion.
  ST-2427: Investigational drug
- Single Ascending Dose: Cohort 4: 22 mg ST-2427 (n=4) administered once over a 60-minute intravenous (IV) infusion.
  ST-2427: Investigational drug
- Pooled Placebo: placebo (n=2 per cohort) administered once over a 60-minute intravenous (IV) infusion.
  Placebo: 5% Dextrose Injection
Period: Overall Study
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Started | 4 | 4 | 4 | 4 | 8
Completed | 4 | 4 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pooled Placebo: Pooled placebo (n=8) administered once over a 60-minute intravenous (IV) infusion.
  Placebo: 5% Dextrose Injection
- Total: Total of all reporting groups
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (6.73) | 49.5 (3.42) | 40.0 (9.93) | 32.5 (13.03) | 43.4 (11.13) | 41.5 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 1 | 3
  Male | 3 | 3 | 4 | 4 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 4 | 4 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4 | 4 | 12
  White | 1 | 4 | 2 | 0 | 3 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: For purposes of monitoring safety, treatment-emergent adverse events (AEs) will be graded using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers (FDA 2007) which is appropriate for healthy subjects.
Time Frame: Day 1 through Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
Participants | 3 | 1 | 2 | 1 | 2

2. Primary Outcome: Number of Participants With Adverse Events Assessed by Blood Pressure
Description: Blood pressure, including orthostatic blood pressure (BP; diastolic blood pressure [DBP], systolic blood pressure [SBP]), will be used to analyze for change from baseline. Adverse events assessed by blood pressure include hypertension and hypotension (MedDRA Preferred Term).
Time Frame: Day 1 through Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
Participants | 1 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events Assessed by ECG
Description: Cardiodynamic evaluation will be performed to evaluate the treatment effects on heart rate-corrected QT interval using the Fridericia (QTcF) corrections.
Time Frame: Day 1 through Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Events Assessed by Clinical Laboratory Assessments
Description: Descriptive statistics will be used to evaluate the treatment effects on clinical laboratory assessments including clinical chemistry, hematology, and urinalysis.
Time Frame: Day 1 through Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Adverse Events Assessed by Body Weight
Description: Body weight (kg) will be assessed for changes relative to baseline.
Time Frame: Day 1 through Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Pharmacokinetics of ST-2427 Concentration in Whole Blood: Cmax
Description: PK modeling will be performed using compartmental methods. The maximum concentration of ST-2427 in whole blood after the ST-2427 infusion in the SAD.
Time Frame: 0-48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL | 206 (26.6) | 364 (51.0) | 551 (131) | 860 (226)

7. Secondary Outcome: Pharmacokinetics of ST-2427 Concentration in Whole Blood: Area Under the Curve
Description: PK modeling will be performed using compartmental methods. The AUC (area under the curve) of ST-2427 in whole blood after the ST-2427 infusion in the SAD.
Time Frame: 0-9 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*h/mL | 706 (111) | 1257 (74.2) | 1990 (132) | 2910 (53.3)

8. Secondary Outcome: Pharmacokinetics of ST-2427 Concentration in Whole Blood: Area Under the Curve
Description: as for outcome 7
Time Frame: 0-25 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng*h/mL | 1044 (141) | 1864 (80.0) | 3003 (126) | 4312 (660)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 8
Description: Adverse events were classified by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), version 23.1.
Arm/Group | Single Ascending Dose: Cohort 1 | Single Ascending Dose: Cohort 2 | Single Ascending Dose: Cohort 3 | Single Ascending Dose: Cohort 4 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 2/4 | 1/4 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Ascending Dose: Cohort 1 (N=4) | Single Ascending Dose: Cohort 2 (N=4) | Single Ascending Dose: Cohort 3 (N=4) | Single Ascending Dose: Cohort 4 (N=4) | Pooled Placebo (N=8)
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Infusion site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT04475198/Prot_SAP_000.pdf